CLINICAL TRIAL: NCT06809491
Title: One-year Recurrence-free Survival of Melanoma Patients Eligible for a Sentinel Lymph Node Biopsy
Acronym: MELASENTI
Status: Active, not recruiting | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, Anne Claire BURSZTEJN, Clinical Professor, Central Hospital, Nancy, France
Other Study IDs: 2024_PI_212
Record Dates: First submitted 2025-01-23; First posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Melanoma, Skin; Adjuvant Treatment
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Melanoma is one of the most aggressive solid cancers, although mortality can be reduced with early treatment. Immunotherapy has transformed the prognosis of this pathology.

The sentinel lymph node technique is used to classify the severity of melanoma. It is proposed for melanomas with a Breslow thickness of 0.8 mm to 1 mm, and recommended for melanomas greater than 1 mm or with ulceration, whatever the Breslow index.

This technique is particularly useful for assessing pathology by detecting the presence of lymph node metastases. Patients with lymph node involvement (micro or macro) are eligible for adjuvant treatment.

The new recommendations suggest adjuvant immunotherapy for stages IIB and IIC (without lymph node involvement assessed by the sentinel lymph node technique). This procedure is widely used at the CHRU de NANCY.

The aim of this study is to demonstrate the value of the sentinel lymph node in assessing the risk of melanoma recurrence at one year (or more).

ELIGIBILITY:
Inclusion Criteria:

Major patient with a melanoma with a Breslow index greater than 0.8mm or ulcerated melanoma, non-metastatic at diagnosis,

Exclusion Criteria:

* Metastatic patient
* Minor patient
* Melanoma with a Breslow index of less than 0.8mm and not ulcerated
* Patient objecting to data collection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed at the CHRU de Nancy or at the ICL between 01/01/2019 and 31/12/2023 and who does not object to the collection of his/her data.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-01-23 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Death or recurrence one year after diagnosis | 1 year
  Death or recurrence one year after diagnosis measured through the one-year reassessment (clinical or radiological evaluation).

SECONDARY OUTCOMES:
Overall survival | 4 years
  To evaluate the overall survival one year after diagnosis in melanoma patients eligible for a sentinel lymph node biopsy.
predictive factors of mortality or recurrence one year after diagnosis | 4 years
  To evaluate the predictive factors of mortality or recurrence one year after diagnosis in melanoma patients eligible for a sentinel lymph node biopsy.
the recurrence-free survival | 4 years
  To evaluate the recurrence-free survival of melanoma patients eligible for a sentinel lymph node biopsy.
complications associated with the sentinel lymph node biopsy | 4 years
  To evaluate the complications associated with the sentinel lymph node biopsy.
recurrence-free survival of patients over 70 years old | 4 years
  To evaluate the recurrence-free survival of patients over 70 years old with melanoma eligible for a sentinel lymph node biopsy.
post-sentinel lymph node biopsy treatments | 4 years
  To describe post-sentinel lymph node biopsy treatments
the tolerance of adjuvant treatment. | 4 years
  To document the tolerance of adjuvant treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Vandœuvre-lès-Nancy, Grand Est, France

IPD SHARING:
Plan to Share IPD: Undecided